CLINICAL TRIAL: NCT01626118
Title: A Phase 3, Randomized, Double-Blind, Multiple-Dose, Parallel-Group, Placebo-Controlled Study of Indomethacin Nanoformulation Capsules for the Treatment of Acute Postoperative Pain After Bunionectomy
Brief Title: Study of Indomethacin Capsules to Treat Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IND3-10-06
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Other Acute Postoperative Pain
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Indomethacin 40 mg TID (Experimental)
  Interventions: Drug: Indomethacin
- Indomethacin 40 mg BID (Experimental)
  Interventions: Drug: Indomethacin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Indomethacin 20 mg TID (Experimental)
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Indomethacin — capsules, 40 mg, TID
  Arms: Indomethacin 40 mg TID
Drug: Indomethacin — capsules, 40 mg, BID
  Arms: Indomethacin 40 mg BID
Drug: Indomethacin — capsules, 20 mg, TID
  Arms: Indomethacin 20 mg TID
Drug: Placebo — capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Indomethacin [Test] Capsules are safe and effective for the treatment of postoperative bunionectomy pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 65 years of age
* For women of child-bearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control
* Has undergone primary, unilateral, first metatarsal bunionectomy with no additional collateral procedures
* Patient must be willing to stay at the study site ≥ 72 hours

Exclusion Criteria:

* Patient has hypersensitivity, allergy, or clinically significant intolerance to any medications to be used in the study, or related drugs
* Patient has a current disease or history of a disease that will impact the study or the patient's well-being
* Patient has used or intends to use any of the medications that are prohibited by the protocol
* Patient has a history of drug or alcohol abuse or dependence, or patient has a positive urine drug screen or alcohol breathalyzer test
* Patient has taken another investigational drug within 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Dickerson, DPM, Principal Investigator — Premier Research Group Limited; Michael Golf, DPM, Principal Investigator — Premier Research Group Limited; Ira Gottlieb, DPM, Principal Investigator — Chesapeake Research Group, LLC; Kyle Patrick, DO, Principal Investigator — Premier Research Group Limited
Locations (4):
- United States (4):
  - Premier Research Group Limited, Phoenix, Arizona
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - Premier Research Group Limited, Austin, Texas
  - Premier Research Group Limited, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Indomethacin 40 mg TID: Indomethacin Nanoformulation Capsules 40 mg TID
- Indomethacin 40 mg BID: Indomethacin Nanoformulation Capsules 40 mg BID
- Indomethacin 20 mg TID: Indomethacin Nanoformulation Capsules 20 mg TID
- Placebo: Placebo Group
Period: Overall Study
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Started | 94 | 93 | 92 | 94
Completed | 92 | 91 | 90 | 91
Not Completed | 2 | 2 | 2 | 3
Not completed — Lack of Efficacy | 1 | 0 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Investigator Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo | Total
Number analyzed (Participants) | 94 | 93 | 92 | 94 | 373
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (12.27) | 38.9 (12.5) | 41.3 (12.57) | 40.7 (11.32) | 40.3 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 77 | 77 | 83 | 317
  Male | 14 | 16 | 15 | 11 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 26 | 12 | 20 | 73
  Not Hispanic or Latino | 79 | 67 | 80 | 74 | 300
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Subjects were allowed to select more than one race; therefore, some subjects are counted multiple times.
  participants
    American Indian or Alaska Native | 2 | 2 | 0 | 1 | 5
    Asian | 2 | 2 | 2 | 2 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 0 | 3
    Black or African American | 15 | 25 | 21 | 19 | 80
    White or Caucasian | 77 | 66 | 69 | 70 | 282
    Other | 0 | 0 | 1 | 2 | 3
Weight (kg) [Mean (Standard Deviation); unit: KG] — Weight measured in kilogram
  KG | 73.81 (14.686) | 72.77 (15.761) | 74.99 (17.821) | 71.22 (14.607) | 73.19 (15.758)
Height (cm) [Mean (Standard Deviation); unit: CM] — Height measured in centimeters
  CM | 166.28 (8.059) | 165.65 (8.994) | 166.52 (9.761) | 165.61 (7.646) | 166.01 (8.621)
BMI (kg/m^2) [Mean (Standard Deviation); unit: KG/M^2] — Body mass index measured in kilograms per meter squared.
  KG/M^2 | 26.5 (4.49) | 26.3 (4.34) | 26.7 (4.73) | 25.8 (4.57) | 26.3 (4.52)
Baseline pain intensity, mm [Mean (Standard Deviation); unit: mm] — The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".
  mm | 71.0 (16.33) | 71.2 (16.11) | 72.3 (15.90) | 73.9 (16.6) | 72.1 (16.21)
Surgery duration, min [Mean (Standard Deviation); unit: minutes] — Surgery duration, minutes
  minutes | 27.7 (7.45) | 27.6 (7.95) | 28.5 (8.63) | 27.2 (6.59) | 27.7 (7.67)

OUTCOME MEASURES:

1. Primary Outcome: The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale From 0 to 48 Hours After Trial Entry (VASSPID-48)
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain". Pain intensity is assessed at baseline (time "0") and at the following time points after time 0: 15, 30, and 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 32, 40, and 48 hours.
  The VAS summed pain intensity difference (VASSPID) is calculated as the sum of the pain intensity difference values at each follow-up time point (difference between the starting pain intensity and the pain intensity at the given assessment time) multiplied by the amount of time (in hours) since the prior assessment.
Time Frame: 0-48 hours
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug.
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Number analyzed (Participants) | 94 | 93 | 92 | 94
mm*hour | 598.670 (1173.7863) | 623.162 (1182.0912) | 342.779 (858.6326) | 280.517 (817.6026)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; The p value was obtained from an analysis of covariance (ANCOVA) model that included treatment effect as the factor and baseline pain intensity as the covariate. This was the primary analysis of the primary efficacy parameter; Test type: Superiority or Other; p = 0.034, ANCOVA; Difference in Least Squares Mean = 317.612, 95% CI 2-sided [23.297 to 611.926], Standard Error of Mean 149.6694
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.023, ANCOVA; Difference in Least Squares Mean = 342.132, 95% CI 2-sided [47.090 to 637.175], Standard Error of Mean 150.0397
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.680, ANCOVA; Difference in Least Squares Mean = 61.972, 95% CI 2-sided [-233.527 to 357.471], Standard Error of Mean 150.2717
Statistical Analysis 4: Comparison: Indomethacin 40 mg TID vs Placebo; The p value was obtained from a mixed-model repeated-measure (MMRM) model that used all available data from all subjects to derive an estimate of pain intensity scores for subjects following study withdrawal, rather than "imputing" a score for individual subjects. The MMRM analysis was a sensitivity analysis of the primary efficacy parameter; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in Least Squares Mean = 503.008, 95% CI 2-sided [301.930 to 704.086], Standard Error of Mean 102.3149
Statistical Analysis 5: Comparison: Indomethacin 40 mg BID vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in Least Squares Mean = 511.357, 95% CI 2-sided [309.749 to 712.965], Standard Error of Mean 102.5851
Statistical Analysis 6: Comparison: Indomethacin 20 mg TID vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in Least Squares Mean = 341.232, 95% CI 2-sided [139.249 to 543.215], Standard Error of Mean 102.7761

2. Secondary Outcome: VASSPID-4. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 4 Hours After Trial Entry.
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain". Pain intensity is assessed at baseline (time "0") and at the following time points after time 0: 15, 30, and 45 minutes and 1, 1.5, 2, 3, and 4 hours.
  The VAS summed pain intensity difference (VASSPID) is calculated as the sum of the pain intensity difference values at each follow-up time point (difference between the starting pain intensity and the pain intensity at the given assessment time) multiplied by the amount of time (in hours) since the prior assessment.
Time Frame: 0-4 hours
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug.
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Number analyzed (Participants) | 94 | 93 | 92 | 94
mm*hour | 31.5 (74.4) | 35.3 (79.6) | 24.8 (54.6) | 18.4 (62.1)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.191, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.108, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.461, t-test, 2 sided

3. Secondary Outcome: VASSPID-8. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 8 Hours After Trial Entry.
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain". Pain intensity is assessed at baseline (time "0") and at the following time points after time 0: 15, 30, and 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 hours.
  The VAS summed pain intensity difference (VASSPID) is calculated as the sum of the pain intensity difference values at each follow-up time point (difference between the starting pain intensity and the pain intensity at the given assessment time) multiplied by the amount of time (in hours) since the prior assessment.
Time Frame: 0-8 hours
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug.
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Number analyzed (Participants) | 94 | 93 | 92 | 94
mm*hour | 69.7 (151.7) | 75.5 (152.5) | 47.6 (109.9) | 35.8 (107.9)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.079, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.041, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.458, t-test, 2 sided

4. Secondary Outcome: VASSPID-24. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 24 Hours After Trial Entry.
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain". Pain intensity is assessed at baseline (time "0") and at the following time points after time 0: 15, 30, and 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, and 24 hours.
  The VAS summed pain intensity difference (VASSPID) is calculated as a time-weighted sum of the pain intensity difference values at each follow-up time point (difference between the starting pain intensity and the pain intensity at the given assessment time) multiplied by the amount of time (in hours) since the prior assessment.
Time Frame: 0-24 hours
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug.
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Number analyzed (Participants) | 94 | 93 | 92 | 94
mm*hour | 268.4 (526.9) | 265.2 (516.2) | 156.8 (384.0) | 115.5 (346.5)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.020, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.021, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.441, t-test, 2 sided

5. Secondary Outcome: Total Pain Relief (TOTPAR) Over 0 to 4 Hours (TOTPAR-4).
Description: Pain relief was assessed with a 5-point categorical scale at all assessment timepoints after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none=0, a little=1, some=2, a lot=3 and complete=4. Pain relief is assessed at the following points after time 0: 15, 30 & 45 minutes and 1, 1.5, 2, 3 & 4 hours.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. Thus, individual scores covering a longer period were given more weight. The minimum theoretical score is 0 units, which represents no pain relief (0 on scale) at all points after time 0. The maximum theoretical score is 16 units, which represents complete pain relief (4 on scale) at all points after 0.
Time Frame: 0-4 hours
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Number analyzed (Participants) | 94 | 93 | 92 | 94
units on a scale*hour | 2.6 (3.8) | 2.8 (3.8) | 2.0 (2.9) | 1.9 (3.1)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.141, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.071, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.716, t-test, 2 sided

6. Secondary Outcome: TOTPAR-8. Total Pain Relief (TOTPAR) Over 0 to 8 Hours
Description: Pain relief was assessed with a 5-point categorical scale at all assessment timepoints after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none=0, a little=1, some=2, a lot=3 and complete=4. Pain relief is assessed at the following points after time 0: 15, 30 & 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7 & 8 hours.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. Thus, individual scores covering a longer period were given more weight. The minimum theoretical score is 0 units, which represents no pain relief (0 on scale) at all points after time 0. The maximum theoretical score is 32 units, which represents complete pain relief (4 on scale) at all points after 0.
Time Frame: 0-8 hours
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug.
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Number analyzed (Participants) | 94 | 93 | 92 | 94
units on a scale*hour | 5.0 (8.0) | 5.4 (8.1) | 3.5 (5.9) | 3.0 (5.8)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.049, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.020, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.593, t-test, 2 sided

7. Secondary Outcome: TOTPAR-24. Total Pain Relief (TOTPAR) Over 0 to 24 Hours
Description: Pain relief was assessed with a 5-point categorical scale at all assessment timepoints after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none=0, a little=1, some=2, a lot=3 and complete=4. Pain relief is assessed at the following points after time 0: 15, 30 & 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, & 24 hours.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. Thus, individual scores covering a longer period were given more weight. The minimum theoretical score is 0 units, which represents no pain relief (0 on scale) at all points after time 0. The maximum theoretical score is 96 units, which represents complete pain relief (4 on scale) at all points after 0.
Time Frame: 0-24 hours
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug.
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Number analyzed (Participants) | 94 | 93 | 92 | 94
units on a scale*hour | 16.2 (29.1) | 16.8 (28.0) | 10.1 (21.8) | 7.8 (19.1)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.021, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.012, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.447, t-test, 2 sided

8. Secondary Outcome: TOTPAR-48. Total Pain Relief (TOTPAR) Over 0 to 48 Hours
Description: Pain relief was assessed with a 5-point categorical scale at all assessment timepoints after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none=0, a little=1, some=2, a lot=3 and complete=4. Pain relief is assessed at the following points after time 0: 15, 30 & 45 minutes and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 32, 40 & 48 hours.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. Thus, individual scores covering a longer period were given more weight. The minimum theoretical score is 0 units, which represents no pain relief (0 on scale) at all points after time 0. The maximum theoretical score is 192 units, which represents complete pain relief (4 on scale) at all points after 0.
Time Frame: 0-48 hours
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug.
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Number analyzed (Participants) | 94 | 93 | 92 | 94
units on a scale*hour | 34.7 (65.1) | 37.0 (64.5) | 21.2 (49.3) | 17.3 (45.6)
Statistical Analysis 1: Comparison: Indomethacin 40 mg TID vs Placebo; Test type: Superiority or Other; p = 0.036, t-test, 2 sided
Statistical Analysis 2: Comparison: Indomethacin 40 mg BID vs Placebo; Test type: Superiority or Other; p = 0.017, t-test, 2 sided
Statistical Analysis 3: Comparison: Indomethacin 20 mg TID vs Placebo; Test type: Superiority or Other; p = 0.577, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Indomethacin 40 mg TID | Indomethacin 40 mg BID | Indomethacin 20 mg TID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/93 | 0/92 | 0/94
Other Adverse Events (participants affected / at risk) | 65/94 | 74/93 | 68/92 | 71/94
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indomethacin 40 mg TID (N=94) | Indomethacin 40 mg BID (N=93) | Indomethacin 20 mg TID (N=92) | Placebo (N=94)
Nausea (Gastrointestinal disorders) | 32 | 36 | 34 | 33
Postprocedural edema (Injury, poisoning and procedural complications) | 20 | 18 | 25 | 29
Dizziness (Nervous system disorders) | 16 | 12 | 12 | 16
Headache (Nervous system disorders) | 17 | 12 | 9 | 14
Vomiting (Gastrointestinal disorders) | 9 | 12 | 11 | 8
Constipation (Gastrointestinal disorders) | 3 | 7 | 8 | 5
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 7 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No